CLINICAL TRIAL: NCT04571424
Title: Phase 1, Randomized, Blinded, Placebo-Controlled, Single-Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Dapirolizumab Pegol (BIIB133) in Healthy Japanese and Caucasian Study Participants
Brief Title: A Study to Evaluate Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of BIIB133 (Dapirolizumab Pegol) in Healthy Japanese and Caucasian Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 253HV101
Record Dates: First submitted 2020-09-25; First posted 2020-10-01 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — dapirolizumab pegol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort 1: BIIB133 Dose 1 (Experimental): Participants will receive single IV infusion of BIIB133 Dose 1.
  Interventions: Drug: BIIB133 (Dapirolizumab pegol)
- Cohort 2: BIIB133 Dose 2 (Experimental): Participants will receive single IV infusion of BIIB133 Dose 2.
  Interventions: Drug: BIIB133 (Dapirolizumab pegol)
- Cohort 1-2: Placebo (Placebo Comparator): Participants will receive single IV infusion of matching placebo to BIIB133.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BIIB133 (Dapirolizumab pegol) — Administered as specified in the treatment arm
  Other Names: DZP
  Arms: Cohort 1: BIIB133 Dose 1; Cohort 2: BIIB133 Dose 2
Drug: Placebo — Administered as specified in the treatment arm
  Arms: Cohort 1-2: Placebo

SUMMARY:
The primary objective of the study is to assess the safety and tolerability of a single intravenous (IV) dose of dapirolizumab pegol (DZP) in Japanese healthy study participants compared with those of Caucasian healthy study participants.

The secondary objectives of the study are to assess the pharmacokinetic(s) (PK) of a single IV dose of DZP in Japanese and Caucasian healthy study participants, to evaluate ethnic sensitivity on the PK of DZP between body weight- and gender-matched Japanese and Caucasian healthy study participants and to evaluate the immunogenicity of a single IV dose of DZP in Japanese and Caucasian healthy study participants.

ELIGIBILITY:
Key Inclusion Criteria:

* Negative polymerase chain reaction (PCR) test result for severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) within 14 days of Day -1 (inclusive).
* Japanese study participant has both biological parents and all 4 grandparents of Japanese descent and, if living outside of Japan for more than 5 years, must maintain a Japanese diet.
* Caucasian study participant has both biological parents and all 4 grandparents of Caucasian descent.
* Have a body weight between 50 and 90 kilograms (kg) (inclusive) and body mass index (BMI) between 18.0 and 26.0 kilograms per meter square (kg/m^2) (inclusive) at the Screening Visit.

Key Exclusion Criteria:

* History of any clinically significant cardiac, endocrine, gastrointestinal, hematologic, hepatic, immunologic, metabolic, urologic, pulmonary, neurologic, dermatologic, psychiatric, or renal disease, or other major disease, as determined by the Investigator.
* Have undergone major surgery in the last 6 months or plans to undergo elective major surgery during the study period.
* Have a known hypersensitivity to any components or excipients of DZP including polyethylene glycol (PEG).
* Have received any prescription or nonprescription medicines including over-the-counter remedies and herbal and dietary supplements within 14 days or 5 half-lives of the respective drug, whichever is longer, other than acetaminophen and antihistamines.
* Current enrollment in any other drug, biological, device, or clinical study, or treatment with an investigational drug or approved therapy for investigational use within 30 days prior to Day -1, or 5 half-lives, whichever is longer.
* History of chronic, recurrent, or recent (within 6 months prior to Screening) severe infection and/or at risk for severe infection, as determined by the Investigator.
* Have symptoms consistent with SARS-CoV-2 infection, per the judgement of the Investigator, within 14 days prior to Day -1, including but not limited to fever (temperature > 37.5 degree Celsius [°C]), sore throat, new and persistent cough, breathlessness, or loss of taste or smell.
* Have close contact within 14 days prior to Day -1 with a SARS-CoV-2 (+) individual. Close contact is defined as (1) being within 6 feet of an infected individual (as confirmed via laboratory assessment) for at least 15 minutes within 2 days of symptom onset or (2) being within 6 feet of an asymptomatic infected individual for at least 15 minutes within 2 days of that asymptomatic individual undergoing specimen collection for SARS-CoV-2 testing.
* Clinically significant abnormal laboratory test result values, as determined by the Investigator, at Screening or Day -1.
* Have received any live/attenuated vaccination within 6 weeks prior to Visit 2 (Day 1) or plans to receive any live/attenuated vaccination within 120 days after the dose of study treatment.

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2020-10-14 (Actual); Primary Completion 2021-04-08 (Actual); Study Completion 2021-04-08 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Treatment-emergent Adverse Events (AEs) and Serious Adverse Events (SAEs) | Up to Day 120
  An AE is any untoward medical occurrence in a participant administered a pharmaceutical product and that does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product. An SAE is any untoward medical occurrence that at any dose results in death, places the participant at immediate risk of death, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, results in a birth defect.

SECONDARY OUTCOMES:
Plasma BIIB133 Concentration | Up to Day 120
Area under Concentration-Time Curve from Time 0 to Infinity (AUCinf) of BIIB133 | Up to Day 120
Area under Concentration-Time Curve from Time 0 to Time t (AUC0-t) of BIIB133 | Up to Day 120
Maximum Observed Concentration (Cmax) of BIIB133 | Up to Day 120
Time to Reach Maximum Observed Concentration (Tmax) of BIIB133 | Up to Day 120
Elimination Half-life (t½) of BIIB133 | Up to Day 120
Clearance (CL) of BIIB133 | Up to Day 120
Volume of Distribution (Vd) of BIIB133 | Up to Day 120
Percentage of AUCinf Obtained by Extrapolation (AUCextr%) of BIIB133 | Up to Day 120
Area under Concentration-Time Curve from Time 0 to Infinity Normalized by Dose (AUCinf/Dose) of BIIB133 | Up to Day 120
Area under Concentration-Time Curve from Time 0 to Time t Normalized by Dose (AUC0-t/Dose) of BIIB133 | Up to Day 120
Maximum Observed Concentration Normalized by Dose (Cmax/Dose) of BIIB133 | Up to Day 120
Plasma Polyethylene Glycol (PEG) Concentration | Up to Day 120
AUCinf of PEG | Up to Day 120
AUC0-t of PEG | Up to Day 120
Cmax of PEG | Up to Day 120
Tmax of PEG | Up to Day 120
t½ of PEG | Up to Day 120
AUCextr% of PEG | Up to Day 120
AUCinf/Dose of PEG | Up to Day 120
AUC0-t/Dose of PEG | Up to Day 120
Cmax/Dose of PEG | Up to Day 120
Urine PEG Concentration | Up to Day 120
Ratio of AUCinf of BIIB133 between Japanese and Caucasian Participants | Up to Day 120
Ratio of AUC0-t of BIIB133 between Japanese and Caucasian Participants | Up to Day 120
Ratio of Cmax of BIIB133 between Japanese and Caucasian Participants | Up to Day 120
Ratio of t½ of BIIB133 between Japanese and Caucasian Participants | Up to Day 120
Ratio of CL of BIIB133 between Japanese and Caucasian Participants | Up to Day 120
Ratio of Vd of BIIB133 between Japanese and Caucasian Participants | Up to Day 120
Ratio of AUCinf/Dose of BIIB133 between Japanese and Caucasian Participants | Up to Day 120
Ratio of AUC0-t/Dose of BIIB133 between Japanese and Caucasian Participants | Up to Day 120
Ratio of Cmax/Dose of BIIB133 between Japanese and Caucasian Participants | Up to Day 120
Number of Participants with Anti-BIIB133 Antibodies | Up to Day 120
Plasma Concentration of Anti-BIIB133 Antibodies | Up to Day 120
Number of Participants with Anti-PEG Antibodies | Up to Day 120
Plasma Concentration of Anti-PEG Antibodies | Up to Day 120

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen; Amina Haggag, M.D, Principal Investigator — Anaheim Clinical Trials
Locations (1):
- Anaheim Clinical Trials, Anaheim, California, United States

IPD SHARING:
Plan to Share IPD: Yes
In accordance with Biogen's Clinical Trial Transparency and Data Sharing Policy on https://www.biogentrialtransparency.com/
URL: https://vivli.org/